CLINICAL TRIAL: NCT04492540
Title: Correlation Between Sex Hormones and Different Functions in Response to Aerobic Exercise and MIND Diet in Older Adult Women
Brief Title: Response of Sex Hormones and Different Functions to Exercise and Diet in Elderly Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, marwa mahmoud elsayed mahmoud, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: P.T.REC/012/002773
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Cognitive Decline; Postmenopausal Disorder
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aerobic exercise and MIND diet program (Other): the aerobic exercise in form of treadmill training intensity of exercise moderate intensity, target heart rate (THR) will be 60-70% of heart maximum (HR MAX), time of session 60 min initial 10 min warm up exercise on treadmill in low intensity and target phase 40 min intensity will increase until patient reach to THR then intensity decrease until session will be ended by cooling down phase for 10 min . The volunteers will perform exercise 3 times per week for 12 weeks
  Interventions: Other: aerobic exercise and MIND diet program
- The Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) diet program (Other): the control group will receive MIND diet program for 12 weeks
  Interventions: Other: MIND diet program

INTERVENTIONS:
Other: aerobic exercise and MIND diet program — the aerobic exercise in form of treadmill training intensity of exercise moderate intensity, target heart rate (THR) will be60-70% of heart maximum (HR MAX), time of session 60 min initial 10 min warm up exercise on treadmill in low intensity and target phase 40 min intensity will increase until patient reach to THR then intensity decrease until session will be ended by cooling down phase for 10 min . The volunteers will perform exercise 3 times per week for 12 weeks
  Arms: aerobic exercise and MIND diet program
Other: MIND diet program — control group will receive diet program for 12 weeks
  Arms: The Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) diet program

SUMMARY:
It is an interventional study in which 60 women estimated to enroll according to random allocation and divided into two groups. The study group will receive aerobic exercise in addition to diet restriction while the control group will receive diet recommendations. the aerobic exercise in form of treadmill training intensity of exercise moderate intensity, target heart rate (THR) will be 50-60% of heart maximum (HR MAX), time of session 40 min initial 10 min warm up exercise on treadmill in low intensity and active phase 20- 30 min intensity will increase until patient reach to THR then intensity decrease until session will be ended by cooling down phase for 10 min . The volunteers will perform exercise 3 times per week for 12 weeks .different functions and markers will be measured and sex hormones (estradiol ,testosterone. sex hormone binding globin ) pre and post

DETAILED DESCRIPTION:
PURPOSE:

to determine the effect of aerobic exercise and diet on sex hormones and different functions and markers, and if is there correlation between two factors effect in postmenopausal elderly women

BACKGROUND:

Alzheimer's disease (AD) is the most common neurodegenerative disease, accounting for more than 50% of all dementia types. Its twice more common in females which could be due to increased longevity and sex difference in brain size .Estrogen has neurotrophic action in areas involved in memory and cognition. Post-menopausal women are at increased risk than their male counterpart. Women with Alzheimer have lower endogenous estrogen level which lead to the hypothesis that estrogen could be neuroprotective. Estrogen and androgen receptors are widely distributed throughout the brain e.g. in the cerebral cortex, amygdala, hypo-thalamus and also in the hippocampus which is important for cognitive functioning. There are shown clear associations between sex hormones and activities in memory, emotional and rewarding circuits in the brain measured with functional magnetic resonance imaging, several significant correlations were found between serum hormone levels and spatial ability. High absolute estrogen levels, a high estrogen/testosterone ratio and increasing levels during estrogen treatment were all associated with lower spatial ability. This is in agreement with many previous reports of sex differences where women in general tend to perform worse than men in this specific aspect of cognitive function. In menstruating women, a deterioration of spatial ability was demonstrated during high levels of circulating estrogen, and it was improved during the menstrual phase of the cycle when hormone levels are lowest.

HYPOTHESES:

There is no correlation between sex hormones and different functions and markers in response to aerobic exercise and diet in elderly postmenopausal women

RESEARCH QUESTION:

Is there correlation between sex hormones and different functions and markers in elderly postmenopausal women in response to aerobic exercise and dietary restriction?

ELIGIBILITY:
Inclusion Criteria:

* • Sixty Postmenopausal women (60-70 y)

  * Body mass index (BMI) ranged from 30 to 39.9 kg/m2

Exclusion Criteria:

* • regular medications(e.g., β-blockers, α-blockers, digoxin, diuretics, aspirin, nitrates, Presently using sex hormones)

  * having active chronic illness (e.g., rheumatoid arthritis, hyperthyroidism, and inflammatory bowel disease) and diabetes mellitus or other (unstable) endocrine-related diseases
  * presence of malignant disease
  * blood donation within the last 30 days
  * Participation as a subject in any type of study or research during the prior 90 days

Ages: 60 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-20 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
sex hormones | 12 weeks
  level of sex hormones(estradiol ,testosterone. sex hormone binding globin )
cognitive functions | 12 weeks
  cognitive functions by Rowland Universal Dementia Assessment Scale(RUDAS)which has a high score of 30 points, where the least scores indicate severe cognitive impairment
functional level | 12 weeks
  measuring functional level by Functional Independence Measure(FIM) it is ranging from 18 (lowest) to 126 (highest) level of independence: Items are scored on a 7-point ordinal scale, with 7 reflecting complete independency and 1 reflecting total dependence. Scores of 1 to 5 indicate a need for caregiver assistance

CONTACTS AND LOCATIONS:
Overall Officials: ghada e Elrefaye, phd, Study Director — physical therapy faculty Cairo university
Locations (1):
- Physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: one year after completing the study
Access Criteria: journal publishes the study
URL: http://Scholar.cu.edu.eg/p_t